CLINICAL TRIAL: NCT06337487
Title: Relevance of Health-related Quality of Life Assessment for Early Identification of Supportive Care Needs in Oncology Patients
Brief Title: Quality of Life Assessment for Early Identification of Supportive Care Needs in Oncology Patients
Acronym: SOS-DETEQT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/716
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Oncology
Keywords: Supportive care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients, nurses and health professionals and professionals assimilated to the health are recruited in 3 different groups but no comparison will be made between them. Recruitment of patients will be stopped once 79 analyzable patients will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients (Experimental): Quality of life and satisfaction assessment
  Interventions: Other: QoL questionnaires; Other: Patients satisfaction survey
- Nurses (Other): Assess the value of nurses using the Quality of Life (QoL) scores from the EORTC QLQ-C30 questionnaire to help identify SOS needs at the start of care.
  Interventions: Other: Qualitative Interview (for one part of nurses only); Other: ORIC questionnaire; Other: Professionals satisfaction survey
- Health professionals and professionals assimilated to the health (Other): ORIC questionnaire
  Interventions: Other: ORIC questionnaire

INTERVENTIONS:
Other: QoL questionnaires — The EORTC QLQ-C30 questionnaire is a specific cancer questionnaire. A score is calculated per dimension reflecting the patient's level for the corresponding QoL scale (dimension). These scores are calculated according to the EORTC recommendations.
  Research work was recently developed by Giesinger et al. within the EORTC QoL group, with the aim of providing thresholds of clinical importance for the different dimensions of the QLQ-C30.
  An item was added to complete the QLQ-C30. It comes from the EORTC bank library item based on the INCa organizational framework. This item was chosen because it addressed a theme not addressed in the QLQ-C30, sexual health. After consultation with a multidisciplinary team, the threshold was determined for this additional item. "Has your illness or treatment had a negative effect on your sex life? ", the threshold is reached when the answer is "enough" or "a lot."
  Arms: Patients
Other: Qualitative Interview (for one part of nurses only) — At the end of the study, semi-directed qualitative interviews will be conducted with the nurses carrying out the TAS with the aim of understanding the obstacles and facilitators of the routine implementation of the QoL assessment to early identify the SOS needs of patients treated in medical oncology. The semi-structured interviews will be accompanied by an interview grid composed of main questions and follow-up questions. The main questions help introduce the theme. The follow-up questions make it possible to clarify the participants' comments without interrupting the fluidity of the exchanges. The themes discussed between the researcher and the participant during the interview will be as follows: Personal information and overall professional experiences, Knowledge of the study and experience of training with tools (questionnaire and software), Perception of tools (questionnaire and software) and their implementation, Definition and perception of key concepts.
  Arms: Nurses
Other: ORIC questionnaire — Organisational readiness is a factor known to influence the predisposition of individuals to change within an organisation. Based on Weiner's organisational theory, Organizational Readiness for Implementing Change (ORIC) is a questionnaire that has been developed and validated, particularly in French, to measure the organisation's state of in the field of healthcare. It comprises ten items which measure two concepts: commitment to change and effectiveness of change.
  Arms: Health professionals and professionals assimilated to the health; Nurses
Other: Professionals satisfaction survey — A satisfaction questionnaire will be offered to all professionals involved once the last patient has been included. This questionnaire has previously been developed by the UMQVC team to assess investigator satisfaction for other studies and adapted to the context of SOS-Deteqt.
  This questionnaire evaluates in particular :
  * the quality of training
  * ease of use of the CHES
  * the relevance of using the CHES and the PROs
  * the relevance of maintaining the PRO evaluation approach in current clinical practice.
  Arms: Nurses
Other: Patients satisfaction survey — A patient satisfaction questionnaire was drawn up for the study. It includes items taken from :
  * the EORTC's PATSAT33 satisfaction questionnaire, and in particular items relating to the quality of information provided by nurses and the time spent
  * the EORTC COMU26 communication evaluation questionnaire, and in particular the items on being comfortable asking questions, professional responses to difficult difficult subjects, explanation of treatment objectives, etc.
  * the questionnaire developed jointly by the UMQVC team and the psychology laboratory of the psychology laboratory at the University of Franche Comté as part of the REMOQOL-Poumon study and assessing in particular
  * understanding of the purpose of using the QoL questionnaire
  * ease of completion and use of the tablet
  * satisfaction with the questionnaire and the tablet
  * intention to use in the future
  Arms: Patients

SUMMARY:
The aim of this study is to evaluate the value of the nurse's use of the Quality of Life (QoL) scores of the European Organisation for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire [QLQ] C30 as an aid in identifying the needs for supportive oncological care at the start of care, in patients followed up for locally advanced or metastatic cancer starting systemic antineoplastic treatment. The main questions it aims to answer are as follows:

* Comparison of the personalised oncology support care plans proposed by the nurse before and after the QoL results were obtained
* The nurse's assessment of the relevance of the information provided by the QOL scores.

During the Care Support Stage (CSS), the nurse will assess the patient's situation during the interview and will fill in directly on an electronic form the Oncological Support Care proposed to the patient, making up the Personalised Pre-QoL Oncological Support Care Plan (PPSOS pre-QoL). The nurse will then give the patient the tablet to fill in the QoL questionnaire. She will then look at the results of the QoL questionnaire and the alerts in the event of deterioration, and will reassess the PPSOS using a new computerised PPSOS post-QoL form. The nurse will assess the relevance of the information provided by the QoL scores concerning the urgency of care, the need to go into certain subjects in greater depth, the identification of problems not addressed before or the discussion of sensitive subjects not addressed before. The nurse will give the patient the tablet to fill in a satisfaction questionnaire. In an attempt to control the biases inherent in an assessment carried out by a single healthcare professional, the clinical records of the patients included will be presented to a group of professionals who will also propose a PPSOS, known as Experts. The group will be made up of a nurse, a medical oncologist and at least two healthcare professionals and professionals in a similar field (dietician, psychologist, APA teacher, social worker, etc.). This group will analyse all the patient files included in the two study centres at dedicated meetings. In order to characterise patient care following the CSS, the oncological support care performed, unscheduled hospitalisations, emergency room visits and calls to the on-call medical team will be collected for the two months following the CSS.

DETAILED DESCRIPTION:
To put in place the conditions needed to move from a "care pathway" centred on the medical management of cancer to a "health pathway" that takes into account all the physical, psychological and social needs of patients and their families.

The incidence of cancer is increasing, due to longer life expectancy and improved diagnostic methods. The announcement of a cancer diagnosis and its treatment have a global and multidimensional impact on patients, so their care should not be limited to the direct symptoms of the disease and the management of the undesirable effects of treatment, but should focus on the person as a whole.

In France, oncological support care (SOS) was defined in the first cancer plan as "all the care and support required by patients throughout their illness, in conjunction with specific onco-haematological treatments, where available". The main aim of SOS is to ensure the best possible Quality of Life (QoL) for the patient. Whether or not they involve medication, they are used in conjunction with specific cancer treatments. It is recommended that SOS needs be identified at the outset of treatment.

The announcement process is a key stage in the care pathway, providing a multi-dimensional assessment of the patient's needs and the impact of the newly diagnosed cancer on his or her environment. There are four stages in this process: a medical stage (announcement and treatment proposal), a healthcare support stage (CSS), access to a team of SOS professionals, and a link-up stage with primary care. The CSS enables an in-depth assessment of the patient's SOS needs.

The use of patient-perceived health data (Patient Reported Outcome, PRO) could help with this assessment by measuring the patient's experience and quantifying the impact of the disease and treatment as experienced directly by the patient. PRO are defined as "any report on the patient's state of health that comes directly from the patient, without interpretation of the patient's response by a clinician or any other person".

QoL is considered to be part of PROs. QoL is a multidimensional and dynamic concept that reflects the patient's perception of the effect of the disease and its treatment on the physical, emotional, functional and social aspects of life in particular.

The oncology methodology and quality of life unit (UMQVC) at the Besançon university hospital centre (CHU) has developed a research project on routine electronic monitoring of the quality of life of patients undergoing cancer treatment: Routine Electronic Monitoring of Quality of Life (REMOQOL). The aim is to use the results of the QOL questionnaire as a complementary tool in the care of patients being monitored for cancer.

As part of this study, the use the PROs is proposed and, more specifically, the QoL assessment, to help identify SOS needs at the start of care. QoL assessment at the start of treatment provides a multidimensional representation of the patient's perceived state of health.

The hypothesis is that the use of the QLQ-C30 QoL questionnaire, with the aid of digital tools, could help with the initial assessment of the SOS needs of patients undergoing medical oncology treatment. This multidimensional assessment will provide a measurable and reproducible value for a measure that can only be assessed directly by the patient.

This initial assessment, during the CSS, could therefore serve as a reference and guide the patient towards specific care pathways, such as referring the patient to a supportive care day hospital, if the patient requires interdisciplinary care. This approach could allow patients to be at the centre of care and encourage their involvement in decision-making.

Ultimately, this questionnaire could be used to help assess patients' needs and monitor their progress at different points in the care process, and could be offered in institutions as well as at home.

ELIGIBILITY:
CRITERIA FOR PATIENTS:

Inclusion Criteria:

* Patient with locally advanced or metastatic cancer
* Patient due to start antineoplastic systemic treatment (immunotherapy, chemotherapy, targeted therapy, etc.) in 1st line,
* Patient able to understand French and fill in questionnaires (no major cognitive impairment),
* Male and female, at least 18 years of age,
* Signature of informed consent to participate, indicating that subject has understood procedures required by the study and that he/she agrees to participate in the study study and to abide by the requirements and restrictions inherent to this study,
* Affiliation with a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Cognitive disorders compromising the comprehension of information or the or completion of QoL questionnaires,
* Patients who were unable to benefit from SBT prior to initiation of their systemic antineoplastic systemic treatment and having already received more than 2 1st-line injections,
* Legal incapacity or limited legal capacity,
* Subject unlikely to cooperate with study and/or poor cooperation anticipated by investigator,
* Subject without health insurance,
* Pregnant woman.

CRITERIA FOR PROFESSIONALS:

For the evaluation of satisfaction and the ORIC questionnaire: all health professionals and professionals assimilated to the health field use the QoL results

For the qualitative analysis: the nurses carrying out the TAS and participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change between pre and post QoL Questionnaires | Day 1
  EORTC QLG Core Questionnaire (EORTC QLQ-C30) + additional item = 31 items submitted to patients.
  Each item of QLQ-C30 is rated from 1 (= not at all) to 4 (= very much). The change between the personalized plan for supportive oncology care completed before the QLQ assessment and the personalized plan for oncology care completed with the graphical results of the QLQ assessment.
  The change is defined by at least one different SOS proposal, regardless of the direction of the difference (addition or removal of an SOS proposal). The pre-QoV PPSOS is drawn up by the nurse after interviewing the patient, without consulting the QoV results. The post-QoV PPSOS is drawn up by the nurse immediately after interviewing the patient, and after reviewing the QoV results via the CHES software.
The nurse's assessement of the relevance of the information provided by each patients's QoL scores | Day1
  The nurse's assessment of the relevance of the information provided by each patient's QoL scores, in terms of the urgency of care, the need for further investigation of certain topics, the identification of issues not previously addressed, or the discussion of sensitive topics not previously addressed. Information will be considered relevant for a patient if at least one of these reasons is mentioned.
  A QoL assessment will be considered as soon as there is a change in the PPSOS and/or relevant information provided by QoL scores.

CONTACTS AND LOCATIONS:
Overall Officials: Magalie Pagnot, Nurse, Principal Investigator — CHU de Besançon
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - Groupement Hospitalier de Haute-Saône, Vesoul

IPD SHARING:
Plan to Share IPD: No